CLINICAL TRIAL: NCT00737646
Title: Evaluation of an Intervention to Increase Colorectal Cancer Screening in Primary Care Clinics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCCDPHP-4555
Record Dates: First submitted 2008-08-15; First posted 2008-08-19 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Colorectal Cancer
Keywords: Cancer; Colorectal cancer; Patient education; Physician education
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms | interventions — Ambulatory Care Facilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Other): Usual care
  Interventions: Behavioral: Usual care
- 2 (Experimental): Clinic-focused intervention: The clinicians and clinical staff in each of the clinics will be scheduled for training sessions. The provider trainings will be designed for clinicians and clinical staff and will be conducted in at least two separate sessions of approximately 3 hours total duration. The sessions will be scheduled to accommodate the clinic schedule, but will be held with no more than 1 month between them. Participants in clinic training sessions will receive continuing education credit.
  Interventions: Behavioral: Clinic-focused intervention
- 3 (Experimental): Clinic-focused and patient focused intervention: The clinic focused-intervention as described in Arm 2 will be combined with a patient-focused intervention.
  Patient focused intervention: CRC education packets, based upon previously developed CDC CRC patient education materials, have been adapted for each study site. These CRC educational packets will be mailed to average-risk patients aged 50-80 years who are due for CRC screening (based on electronic records) and who schedule a non-acute ambulatory care visit in clinics assigned to the patient-focused intervention. A cover letter signed by the patient's physician will be included with each packet. The packets will be mailed approximately 1 week before the medical appointment.
  Interventions: Behavioral: Clinic- and patient-focused

INTERVENTIONS:
Behavioral: Usual care — No intervention will be conducted in this arm of the study.
  Arms: 1
Behavioral: Clinic-focused intervention — The clinic-focused intervention consists of CRC screening training sessions for clinicians and clinical staff. The provider training sessions will include the presentation of CRC screening statistics and information, and will be heavily interactive and skills-based. The provider training sessions will also focus on the provision of tools for improving clinical staff- and clinician-patient interactions about CRC screening and for office system changes/improvements to identify eligible patients and to track screening.
  Arms: 2
Behavioral: Clinic- and patient-focused — This arm will combine the clinic-focused intervention and the patient-focused intervention. The clinic-focused intervention consists of CRC screening training sessions for clinicians and clinical staff as described in Arm 2. The patient-focused intervention includes sending a CRC screening education packet (CDC-developed educational text tailored for use within the study sites), accompanied by a letter from the patient's physician, to patients meeting study inclusion criteria.
  Arms: 3

SUMMARY:
This study is a three-arm randomized controlled trial to implement and evaluate the relative effects of: 1) clinic-focused intervention; 2) combined patient- and clinic-focused intervention, and 3) usual care on the provision of colorectal cancer (CRC) screening in primary care clinics. The study will also examine the relative effects of the intervention conditions on secondary behavioral outcomes (e.g., clinician-patient discussions about CRC screening) and on intermediate outcome measures of attitudes, beliefs, opinions, and social influence surrounding CRC screening among patients, clinicians, and clinical staff. The target population includes average-risk patients aged 50-75 years, clinicians, and clinical staff within the primary care setting. The intervention will be implemented within primary care clinics in two managed care organizations (MCOs). The intervention targets the following CRC screening modalities: fecal occult blood test (FOBT), flexible sigmoidoscopy, colonoscopy, and double contrast barium enema.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for the Patient-focused Intervention

* Average risk
* Male or female
* 50-75 years
* Scheduled for non-acute ambulatory care visit at one of the study sites
* Due for CRC screening including no record of FOBT in the past year, no record of flexible sigmoidoscopy in the past 5 years, no record of colonoscopy in the past 10 years, and no record of double contrast barium enema in the past 5 years

Inclusion Criteria for the Clinic-focused Intervention

* Primary care clinicians, to include the following specialties: Family Practice/General Practice Physicians, General Internal Medicine Physicians, Nurse Practitioners in Family/General Practice, Physician Assistants who conduct non-acute ambulatory medical exams in study clinics
* Primary care clinical staff, to include nurses, medical assistants, and appointment schedulers

Exclusion Criteria (Patients):

* Prior diagnosis of CRC
* Prior diagnosis of colorectal polyps
* Prior diagnosis of ulcerative colitis
* Prior diagnosis of Crohn's Disease
* Prior diagnosis of hereditary nonpolyposis or polyposis
* Medical records contain an International Classification of Diseases (ICD-9) code for family history of CRC
* Younger than 50 years of age
* Older than 80 years of age.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5066 (Actual)
Dates: Start 2009-07; Primary Completion 2010-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Changes in colorectal cancer screening rates (4 modalities) | One year post initiation of intervention

SECONDARY OUTCOMES:
Changes in the frequency of secondary behavioral outcomes (e.g., clinician-patient discussions about CRC screening) | One year post initiation in intervention
Changes in measures of attitudes, beliefs, opinions, and social influence surrounding CRC screening among patients, clinicians, and clinical staff. | One year post initiation of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Judith Lee Smith, PhD, Principal Investigator — Centers for Disease Control and Prevention
Locations (3):
- United States (3):
  - Henry Ford Health System, Detroit, Michigan
  - ABQ Health Partners/Lovelace Clinic Foundation, Albuquerque, New Mexico
  - Battelle Centers for Public Health Research and Evaluation, Seattle, Washington

REFERENCES:
- [Background] Coughlin SS, Costanza ME, Fernandez ME, Glanz K, Lee JW, Smith SA, Stroud L, Tessaro I, Westfall JM, Weissfeld JL, Blumenthal DS. CDC-funded intervention research aimed at promoting colorectal cancer screening in communities. Cancer. 2006 Sep 1;107(5 Suppl):1196-204. doi: 10.1002/cncr.22017. PMID 16802326
- [Background] Shires DA, Divine G, Schum M, Gunter MJ, Baumer DL, Kasprzyk D, Montano DE, Smith JL, Elston-Lafata J. Colorectal cancer screening use among insured primary care patients. Am J Manag Care. 2011;17(7):480-8. PMID 21819168